CLINICAL TRIAL: NCT04247373
Title: The MEC90 of Epidural Ropivacaine Blunting Hemodynamic Changes to Pneumoperitoneum in the Patients Undergoing Laparoscopic Gastrectomy
Brief Title: The MEC90 of Epidural Ropivacaine Blunting Hemodynamic Changes to Pneumoperitoneum
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Jiwon Lee, assistant professor, Keimyung University Dongsan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018-12-036
Record Dates: First submitted 2020-01-23; First posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Laparoscopic Gastrectomy
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- laparoscopic gastrectomy with pneumoperitoneum (Experimental)
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — According to previous patient's response, the investigators will allocate the concentration of ropivacaine of next patient during Co2 insufflation. And, for this allocation of concentration of ropivacaine the investigators use biased coin design up-and-down method.

SUMMARY:
Investigators want to find the concentration of epidural ropivacaine, which can block hemodynamic changes in the onset of pneumoperitoneum in the laparoscopic gastrectomy.

DETAILED DESCRIPTION:
According to previous patient's response, the investigators will allocate the concentration of ropivacaine of next patient during Co2 insufflation. And, for this allocation of concentration of ropivacaine, the investigators use biased coin design up-and-down method.

Based on the practices, the starting concentration is 0.375 %, and the step size of concentration is 0.125%.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing laparoscopic gastrectomy that require pneumoperitoneum
* patients who has epidural catheter to manage postoperative pain control
* patients who agree to our study

Exclusion Criteria:

* patients who don't agree to our study
* BMI<16.0 or BMI>35
* cardiovascular disease, pulmonary disease, renal disease
* alcoholic abuser or drug abuser
* any use of local anesthetics or drugs which have an influence on cardiovascular system from beginning of induction

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in heart rate (bpm) after CO2 insufflation | immediately after CO2 insufflation : 1,2,3,4,5,6, 7, 8, 9, 10 minutes after CO2 insufflation
  Heart rate will be recorded before anesthesia induction, during CO2 insufflation, after Co2 insufflation. The mean value of heart rate before anesthesia induction will be regarded as the baseline values. If maximum heart rate after Co2 insufflation increased by >20% from baseline value, the response will be regarded as "fail" and increased concentration of ropivacaine will be applied to next patient by up and down method.
Changes from baseline in mean arterial pressure (mmHg) after CO2 | immediately after CO2 insufflation : 1,2,3,4,5,6, 7, 8, 9, 10 minutes after CO2 insufflation
  Mean arterial pressure will be recorded before anesthesia induction, during CO2 insufflation, after Co2 insufflation. The mean value of mean arterial pressure before anesthesia induction will be regarded as the baseline values. If maximum mean arterial pressure after Co2 insufflation increased by >20% from baseline value, the response will be regarded as "fail" and increased concentration of ropivacaine will be applied to next patient by up and down method.

CONTACTS AND LOCATIONS:
Overall Officials: JIWON LEE, Dr, Principal Investigator — Dongsan Medical Center